CLINICAL TRIAL: NCT07093996
Title: Endoscopic Pancreatic Duct Stent Placement Versus Conventional Approach in the Treatment of Early Phase Acute Pancreatitis: International Multicenter Controlled Randomized Prospective Study Protocol
Brief Title: Endoscopic Pancreatic Duct Stent Placement Versus Conventional Approach in the Treatment of Early Phase Acute Pancreatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Almazov National Medical Research Centre (Other)
Responsible Party: Principal Investigator, Kotkov Pavel, MD, associate professor of the General Surgery Department Almazov National Medical Research Centre, Almazov National Medical Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14061979
Record Dates: First submitted 2025-07-06; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Acute Pancreatitis (AP)
Keywords: acute pancreatitis; endoscopic pancreatic duct stent placement; pancreatic necrosis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial Masking: not provided (open allocation). Given the specific nature of the medical discipline being studied, blinding of participants, as well as allocation concealment, is not planned due to the practical impossibility of this procedures.
  Randomization method: calendar, according to which patients born in an even year will be distributed into the study group, and those born in an odd year - into the comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Сomparison group (Active Comparator): Treatment measures will be performed in accordance with clinical guidelines and will include infusion therapy, pain relief, and nutritional support. Surgical interventions will also be performed based on estimated indications.
  Interventions: Drug: Conventional treatment of acute pancreatitis in early phase
- Study group (Experimental): Along with the generally accepted complex of therapeutic measures, endoscopic pancreatic duct stent placement will be performed
  Interventions: Procedure: Endoscopic pancreatic duct stent placement

INTERVENTIONS:
Procedure: Endoscopic pancreatic duct stent placement — Endoscopic pancreatic duct stent placement will be performed with a 5Fr Boston Scientific pancreatic stent (3-4 cm in length) within 24 hours from the randomization procedure. The stent will be removed on the 5th day after installation.
  Other Names: Wirsung stenting
  Arms: Study group
Drug: Conventional treatment of acute pancreatitis in early phase — Infusion therapy, pain relief, nutritional support and surgical procedure if needed
  Other Names: Conservative treatment
  Arms: Сomparison group

SUMMARY:
The planned multicenter randomized study is aimed to assess the efficacy and safety of endoscopic pancreatic duct stenting in adult patients with acute pancreatitis. It is planned to include patients with early-stage nonbiliary pancreatitis in the study.

DETAILED DESCRIPTION:
Endoscopic pancreatic duct stent placement is used to treat a variety of pancreatic diseases, including chronic pancreatitis, Wirsung duct strictures, pseudocysts in disconnected duct syndrome and as a preventive measure after endoscopic retrograde cholangiopancreatography. Despite the obvious progress, the greatest number of unsolved problems remain in the issues of using this manipulation in patients with acute pancreatitis. In particular, the perspectives of the pancreatic duct stent placement in treatment of acute pancreatitis early stages remain controversial.

On the one hand, the installation of a stent in the early acute pancreatitis stages helps to normalize the outflow of pancreatic juice from the pancreas and reduce intraductal pressure, leading to a beneficial effect, as evidenced by a number of researchers. On the other hand, stent placement may partially block the second-order pancreatic ducts or increase the risk of sterile pancreatitis contamination due to the development of reflux. In addition, one should not forget about a number of post-manipulation complications inherent in this procedure, including bleeding from the area of the major duodenal papilla, perforation of the duodenum, progression of pancreatic necrosis and cholangitis. Finally, the timing and indications for early endoscopic stenting of the pancreatic duct are not currently standardized, largely due to the fact that acute pancreatitis is a pathological condition that is difficult to predict.

Thus, although this manipulation seems perspective, due to the lack of evidence base, it is currently difficult to recommend it for use in wide clinical practice.

The planned multicenter randomized study is aimed to assess the efficacy and safety of endoscopic pancreatic duct stenting in adult patients with acute pancreatitis. It is planned to include patients with early-stage nonbiliary pancreatitis in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute pancreatitis confirmed on the basis of at least 2 of the 3 diagnostic criteria according to the revised Atlanta classification
2. Presence of organ failure signs (moderate and severe pancreatitis)
3. Informed consent of the patient

Exclusion Criteria:

1. Presence of other indications for endoscopic intervention on the major duodenal papilla (biliary pancreatitis with cholangitis, calculus of the major duodenal papilla, stenosis of the major duodenal papilla, etc.)
2. Previous surgical interventions on the major duodenal papilla
3. Diverticula of the major duodenal papilla
4. Pregnancy
5. Shock
6. Coagulopathy (INR>1.5, blood platelets < 50*109/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | From enrollment to the end of treatment at 3 months
  Data will be tabulated and statistically analyzed in terms of percentages

SECONDARY OUTCOMES:
Incidence of complications associated with endoscopic pancreatic duct stent placement | From endoscopic pancreatic duct stent placement to 3 months
  Frequency of duodenal bleeding, duodenal perforation, unsuccessful major duodenal papilla canulation etc. Data will be tabulated and statistically analyzed in terms of percentages
Rate of different pancreatic necrosis models | From enrollment to the 7th day of treatment
  Will be evaluated according CT-imaging:
  Model 1 - volume of pancreatic necrosis < 30%, or not determined Model 2 - volume of pancreatic necrosis 30-50%, located in the distal pancreatic part Model 3 - volume of pancreatic necrosis 30-50% located in the proximal part Model 4 - volume of pancreatic necrosis 30-50% and more with separation of viable proximal and distal parts (disconnected duct syndrome) Data will be tabulated and statistically analyzed in terms of percentages
Average Balthazar computed tomography severity index (0-10) | From enrollment to the 7th day of treatment
  A scoring system used to assess the severity of acute pancreatitis based on computed tomography scans. Data will be tabulated and statistically analyzed in terms of mean.
Average SOFA (Sequential Organ Failure Assessment Score) score (0-24) | From enrollment to the 7th day of treatment
  Sequential Organ Failure Assessment Score. Data will be tabulated and statistically analyzed in terms of mean
Incidence of other surgical interventions | From enrollment to the end of treatment at 3 months
  Frequency of other surgical interventions, such as abdominal drainage, retroperitoneal drainage, lumbotomy, laparotomy. Data will be tabulated and statistically analyzed in terms of percentages
Number of participants with other surgical interventions | From enrollment to the end of treatment at 3 months
  Number of other surgical interventions, such as abdominal drainage, retroperitoneal drainage, lumbotomy, laparotomy
Length of hospital stay | From date of hospitalization until the date of discharge, assessed up to 3 months
  Data will be tabulated and statistically analyzed in terms of length of hospital stay in days
Number of participants with manifestation of diabetes mellitus | From enrollment to the end of treatment at 3 months
  Data will be tabulated and statistically analyzed in terms of percentages

CONTACTS AND LOCATIONS:
Overall Officials: Badri V Sigua, PhD, Principal Investigator — Almazov National Medical Research Centre
Locations (7):
- Department of General Surgery, Sir Run Run Shaw Hospital, Hangzhou, China
- Russia (6):
  - City Clinical Hospital No. 4, Perm
  - Almazov National Medical Research Centre, Saint Petersburg
  - The City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - I.I. Dzhanelidze research institute of emergency medicine, Saint Petersburg
  - Mariinskaya Hospital, Saint Petersburg
  - Volgograd State Medical University, Volgograd

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leppaniemi A, Tolonen M, Tarasconi A, Segovia-Lohse H, Gamberini E, Kirkpatrick AW, Ball CG, Parry N, Sartelli M, Wolbrink D, van Goor H, Baiocchi G, Ansaloni L, Biffl W, Coccolini F, Di Saverio S, Kluger Y, Moore E, Catena F. 2019 WSES guidelines for the management of severe acute pancreatitis. World J Emerg Surg. 2019 Jun 13;14:27. doi: 10.1186/s13017-019-0247-0. eCollection 2019. PMID 31210778
- [Background] ASGE Standards of Practice Committee; Anderson MA, Fisher L, Jain R, Evans JA, Appalaneni V, Ben-Menachem T, Cash BD, Decker GA, Early DS, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Ikenberry SO, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Shergill AK, Dominitz JA. Complications of ERCP. Gastrointest Endosc. 2012 Mar;75(3):467-73. doi: 10.1016/j.gie.2011.07.010. No abstract available. PMID 22341094